CLINICAL TRIAL: NCT06213792
Title: Visuo-Vestibular Adaptation in Virtual Reality
Acronym: VIVRA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1326
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Healthy Person
Keywords: Vestibulo-Ocular Reflex; Adaptation; Head Impulse Test; Virtual Reality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adaptation of the VOR — Subjects will undergo adaptation of their VOR in virtual reality in two different conditions. The side on which the adaptation will take place and the type of condition with which the patients will start will be randomized. Subject will undergo passive rapid head movements done by an experienced examinator whilst fixing a target in front of them. The movement of the target relative to the movement of the head will increase every 90 seconds by 10% until the movement of the visual scene is twice that of the head movement. In one condition the visual scene will be only a target in a grey void. In the other condition the visual scene will be more complex and represent a target in the room in which the subject is seated. Subjects will undergo both conditions at least 7 days apart.

SUMMARY:
The vestibulo-ocular reflex (VOR) stabilizes the gaze during rapid head movements by inducing an eye rotation of equivalent amplitude but in the opposite direction to the head rotation. Normally, the ratio of eye rotation amplitude to head rotation, or VOR gain, is 1. Under some conditions such as growth or the use of corrective glasses, this gain is adapted to the new visuo-vestibular conditions. This well-known sensorimotor adaptation phenomenon can be achieved through the experimental creation of a conflict between vestibular and visual information.

Incremental velocity error (IVE) allows for a rapid adaption of the VOR at high speed by synchronously projecting a laser target that moves to create a progressively increasing visuo-vestibular conflict. However, this method does not correspond to the ecological conditions of VOR use, as the training is conducted in darkness and the visuo-vestibular conflict does not involve the entire visual scene.

Recreating this type of adaptation in a virtual reality environment could allow for adaptation with a visual stimulus involving the entire visual scene, thus more closely resembling the physiological conditions of VOR use. We hypothesize that a visual simulation of the entire scene would be more effective than an isolated target in VOR adaptation during high velocity head rotation.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 60
* Understanding of the experimental instructions
* Informed Consent

Exclusion Criteria:

* Underlying ENT or neurological disorders
* Corrected Visual Acuity lower than 5/10
* Other conditions leading to oscillopsia or ataxia
* Oculomotor palsy, ocular instability in primary position
* Treatment that may affect ocular motility (psychotropes)
* Cervical rachis pathology with instability
* Cochlear Implants
* Non-stabilized medical disease
* Subject suffering from debilitating motion sickness or Virtual Reality sickness
* Pregnant women
* Patients under tutelage
* Patient without social security

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
VOR gain | 7 days
  VOR gain corresponds to the amplitude of the eye rotation devided by the amplitude of the head rotation for a given head impulse.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Neurologique, Bron, France

IPD SHARING:
Plan to Share IPD: No